CLINICAL TRIAL: NCT00164333
Title: The Treatment Advocacy Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3797; R 18/CCR520972-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: TAP: Treatment Advocacy Program

SUMMARY:
The purpose of the study is to test the efficacy of TAP, a behavioral intervention, in improving sexual safety and treatment adherence among gay and bisexual men infected with HIV. It is hypothesized that those who are in the intervention group will report reductions in unprotected sex with HIV-negative and unknown-status partners; and will show stricter adherence to their treatment regimens, compared to the individuals in the standard-of-care, control group.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ men who have sex with other men, age 18 or over, in HIV care at one of the collaborating clinics, any sexual contact within the previous six months.

Exclusion Criteria:

* self-reported low likelihood of remaining in treatment or in the study location for 12 months, inability to comprehend the consent quiz administered during the Consent and Enrollment Visit, or unwilling to provide required locator information

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09; Primary Completion 2007-05 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Self-reported, unprotected (without condoms) anal or vaginal sex with HIV-negative or unknown-status partners.

SECONDARY OUTCOMES:
Self-reported incidences of missed doses of treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Dogan Eroglu, PhD., Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Howard Brown Medical Center, Chicago, Illinois, United States